CLINICAL TRIAL: NCT00824408
Title: A Randomised Open-label Phase II Trial of BI 6727 Monotherapy and BI 6727 in Combination With Standard Dose Pemetrexed Compared to Pemetrexed Monotherapy in Second Line Non-small Cell Lung Cancer
Brief Title: Trial of BI 6727 (Volasertib) Monotherapy and BI 6727 in Combination With Pemetrexed Compared to Pemetrexed Monotherapy in Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230.5
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; BI 6727

ARMS (2):
- BI 6727 +pemetrexed (Experimental): BI 6727 plus 500 mg/^m2 pemetrexed i.v. on day 1 of 21 day cycle
  Interventions: Drug: pemetrexed; Drug: BI 6727
- pemetrexed (Active Comparator): 500 mg/m^2 i.v. on day 1 of a 21 day cycle
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m^2 i.v. on day 1 of 21 day cycle
  Arms: BI 6727 +pemetrexed
Drug: pemetrexed — 500 mg/m^2 i.v. on day 1 of 21 day cycle
  Arms: pemetrexed
Drug: BI 6727 — BI 6727 i.v. on day 1 of a 21 day cycle
  Arms: BI 6727 +pemetrexed

SUMMARY:
The trial objective will be to evaluate whether BI 6727 monotherapy or in combination with pemetrexed may be effective in the treatment of advanced or metastatic NSCLC in patients who relapsed after or failed first-line platinum based therapy.

The secondary objectives are to identify the acceptable dose of BI 6727 in combination with pemetrexed and to characterize the pharmacokinetic profiles of BI 6727 alone. Arm A, BI6727 monotherapy arm is closed to further recruitment.

ELIGIBILITY:
Inclusion criteria:

1. Pathologic or cytologic confirmed diagnosis of NSCLC
2. Recurrent, advanced or metastatic NSCLC that has progressed following one prior platinum based chemotherapy regimen (not counting adjuvant or neoadjuvant chemotherapy if completed more than 12 months prior to platinum based therapy)
3. Patients who are eligible for pemetrexed as second line chemotherapy
4. Measurable disease by one or more techniques (CT, MRI) according to RECIST
5. Patients aged 18 years or older
6. Life expectancy of at least three (3) months
7. Eastern Cooperative Oncology Group (ECOG) performance Score 0-2
8. Written informed consent that is consistent with ICH-GCP guidelines and local legislation

Exclusion criteria:

1. Treatment with an investigational drug in another clinical study within the past 28 days prior to the start of therapy or concomitantly with this study
2. Anti-cancer therapy for NSCLC (except radiotherapy for palliative reasons) within the past 28 days prior to Treatment Day 1 of Cycle 1 of this trial
3. Any persisting toxicities which are deemed to be clinically significant from the previous therapy
4. Patients who have received more than one prior chemotherapy regimen for advanced disease (not including prior adjuvant therapy). Patients may have received prior epidermal growth factor receptor tyrosine kinase inhibitors.
5. Patients who are unwilling or unable to take folic acid and vitamin B12 supplementation
6. Active brain metastases (stable for <28 days, symptomatic, or requiring concurrent steroids). Patients who have received prior whole brain irradiation and whose brain metastases are stable according to the criteria above will not be excluded.
7. Other active malignancy diagnosed within the past 3 years (other than non melanomatous skin cancer and cervical intraepithelial neoplasia)
8. Concomitant intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would limit compliance with trial requirement or which are considered relevant for the evaluation of the efficacy or safety of the trial drug
9. Patients unable or unwilling to interrupt concomitant administration of NSAIDS 5 days prior to, the day of and 2 days after the administration of pemetrexed, with the exception of lose dose aspirin 81mg daily
10. Patients who have received prior therapy with pemetrexed
11. Absolute neutrophil count (ANC) less than 1,500/mm3
12. Platelet count less than 100,000/mm3
13. Hemoglobin <90g/L
14. Total bilirubin >26µmol/L
15. Alanine amino transferase (ALT) and/or aspartate amino transferase (AST) less than 2.5 X ULN, except in case of known liver metastasis where maximum 5 X ULN is acceptable
16. Serum creatinine level >133µmol/L and/or creatinine clearance (measured or calculated) <45 ml/min
17. Clinically relevant QTc prolongation
18. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
19. Pregnancy or breast feeding
20. Known or suspected active alcohol or drug abuse
21. Patients unable to comply with the protocol
22. Any known hypersensitivity to the trial drugs or their excipients
23. Patients with NSCLC of confirmed Squamous histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Canada (11):
  - 1230.5.00104 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1230.5.00114 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 1230.5.00109 Boehringer Ingelheim Investigational Site, Surrey, British Columbia
  - 1230.5.00107 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1230.5.00105 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1230.5.00119 Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - 1230.5.00116 Boehringer Ingelheim Investigational Site, Oshawa, Ontario
  - 1230.5.00108 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1230.5.00110 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1230.5.00102 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1230.5.00106 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- 1230.5.00118 Boehringer Ingelheim Investigational Site, Nassau, The Bahamas

REFERENCES:
- [Derived] Ellis PM, Leighl NB, Hirsh V, Reaume MN, Blais N, Wierzbicki R, Sadrolhefazi B, Gu Y, Liu D, Pilz K, Chu Q. A Randomized, Open-Label Phase II Trial of Volasertib as Monotherapy and in Combination With Standard-Dose Pemetrexed Compared With Pemetrexed Monotherapy in Second-Line Treatment for Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2015 Nov;16(6):457-65. doi: 10.1016/j.cllc.2015.05.010. Epub 2015 Jun 2. PMID 26100229

RESULTS

PARTICIPANT FLOW:
Groups:
- Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2: Patients received Volasertib 250 mg and pemetrexed 500 mg/m2 administered intravenously (i.v.) on day 1 of each 21 day cycle.
- Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2: Patients received Volasertib 300 mg and pemetrexed 500 mg/m2 administered intravenously (i.v.) on day 1 of each 21 day cycle
- Randomized Phase: Volasertib 300 mg: Patients received Volasertib 300 mg administered intravenously on day 1 of each 21 day cycle
- Randomized Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2: Patients received Volasertib 300 mg and Pemetrexed 500 mg/m2 intravenously on day 1 of each 21 day cycle
- Randomized Phase: Pemetrexed 500 mg/m2: Patients received Pemetrexed 500 mg/m2 administered intravenously (i.v.) on day 1 of each 21 day cycle
Period: Run-in Phase
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomized Phase: Volasertib 300 mg | Randomized Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomized Phase: Pemetrexed 500 mg/m2
Started | 6 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 0 | 0 | 0
Not completed — Progressive disease | 4 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Refused to continue medication | 1 | 0 | 0 | 0 | 0
Not completed — Other reason not defined above | 0 | 1 | 0 | 0 | 0
Period: Randomized Phase
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomized Phase: Volasertib 300 mg | Randomized Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomized Phase: Pemetrexed 500 mg/m2
Started | 0 | 0 | 37 | 47 | 47
Completed | 0 | 0 | 1 (On-treatment at data cutoff (21Dec2012)) | 1 (On-treatment at data cutoff (21Dec2012)) | 1 (On-treatment at data cutoff (21Dec2012))
Not Completed | 0 | 0 | 36 | 46 | 46
Not completed — Not treated | 0 | 0 | 1 | 1 | 1
Not completed — Progressive disease | 0 | 0 | 25 | 36 | 34
Not completed — Adverse Event | 0 | 0 | 4 | 5 | 5
Not completed — Refused to continue medication | 0 | 0 | 2 | 2 | 2
Not completed — Other reason not defined above | 0 | 0 | 4 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Randomized set, which included all patients randomised in the randomisation phase, whether treated or not
Groups:
- Randomization Phase: Volasertib 300 mg: Patients received Volasertib 300 mg administered intravenously (i.v.) on day 1 of each 21 day cycle
- Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2: Patients received Volasertib 300 mg and Pemetrexed 500 mg/m2 intravenously (i.v.) on day 1 of each 21 day cycle
- Randomization Phase: Pemetrexed 500 mg/m2: Patients received Pemetrexed 500 mg/m2 administered intravenously (i.v.) on day 1 of each 21 day cycle
- Total: Total of all reporting groups
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2 | Total
Number analyzed (Participants) | 6 | 6 | 37 | 47 | 47 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.30) | 62.3 (6.83) | 62.9 (8.60) | 63.5 (10.26) | 62.5 (8.89) | 63.1 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 16 | 23 | 25 | 73
  Male | 1 | 2 | 21 | 24 | 22 | 70

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Time From the Date of Randomization to Date of Disease Progression or Death, Whichever Occurred First.
Description: Disease progression was defined according to the Response Evaluation Criteria in Solid Tumours (RECIST)) criteria. Progression-free survival time was calculated as the duration from the date of randomization to the date of disease progression or death, whichever occured first. For patients with known date of progression (or death): PFS [days] = min (date of progression, date of death) - date of randomization + 1 day. For patients without progression or death, PFS was censored at the last imaging date that showed no disease progression: PFS [days, censored] = date of last imaging showing no progression - date randomization + 1 day.
  The number of participants analysed displays the number of patients with an event (progression).
Time Frame: From randomization until disease progression or death
Population: Randomized phase II set, which included all patients who were randomized as part of phase II of the study (not the run in phase)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Number analyzed (Participants) | 34 | 43 | 39
months | 1.4 [1.2 to 1.9] | 3.3 [1.9 to 5.7] | 5.3 [3.1 to 7.2]
Statistical Analysis 1: Comparison: Randomization Phase: Volasertib 300 mg vs Randomization Phase: Pemetrexed 500 mg/m2; Hazard ratio and 95% confidence interval (CI) from Cox proportional-hazards regression model, stratified by histology (Nonsquamous vs. NOS). P-value from log-rank test stratified by histology (one-sided for volasertib 300 mg + pemetrexed 500 mg/m2 vs. pemetrexed 500 mg; two-sided for volasertib 300 mg vs. pemetrexed 500 mg/m2); Test type: Superiority or Other; p = 0.0030, Log Rank; Hazard Ratio (HR) = 2.045, 95% CI 2-sided [1.271 to 3.292]
Statistical Analysis 2: Comparison: Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 vs Randomization Phase: Pemetrexed 500 mg/m2; Hazard ratio and 95% CI from Cox proportional-hazards regression model, stratified by histology (Nonsquamous vs. NOS). P-value from log-rank test stratified by histology (one-sided for volasertib 300 mg + pemetrexed 500 mg/m2 vs. pemetrexed 500 mg/m2; two-sided for volasertib 300 mg vs. pemetrexed 500 mg/m2); Test type: Superiority or Other; p = 0.2804, Log Rank; Hazard Ratio (HR) = 1.141, 95% CI 2-sided [0.735 to 1.771]

2. Secondary Outcome: Objective Tumor Response, Defined as Complete Response (CR), and Partial Response (PR), Evaluated According to RECIST Criteria.
Description: Objective tumor response, defined as complete response (CR), and partial response (PR), evaluated according to RECIST criteria. Evaluation of target lesions: Complete Response (CR): disappearance of all target lesions. Partial Response (PR): ≥30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Evaluation of nontarget lesions: Complete Response (CR): disappearance of all nontarget lesions.
Time Frame: From first drug infusion until 21 days after last drug infusion, up to 1100 days
Population: Randomized set
Measure: Number; unit: percentage of participants
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Number analyzed (Participants) | 6 | 6 | 37 | 47 | 47
percentage of participants
  Complete response (CR) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Partial response (PR) | 16.7 | 50.0 | 8.1 | 21.3 | 10.6
Statistical Analysis 1: Comparison: Randomization Phase: Volasertib 300 mg vs Randomization Phase: Pemetrexed 500 mg/m2; Test type: Superiority or Other; p > 0.9999, Fisher Exact
Statistical Analysis 2: Comparison: Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 vs Randomization Phase: Pemetrexed 500 mg/m2; Test type: Superiority or Other; p = 0.2596, Fisher Exact

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the duration of time from randomization to time of death.
Time Frame: From randomization until time of death
Population: Randomized phase II set, including only patients who died.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Number analyzed (Participants) | 13 | 24 | 23
months | 22.9 [3.6 to NA] — Not calculable due to insufficient data | 17.1 [9.4 to 28.8] | 17.4 [10.3 to 34.6]
Statistical Analysis 1: Comparison: Randomization Phase: Volasertib 300 mg vs Randomization Phase: Pemetrexed 500 mg/m2; Test type: Superiority or Other; p = 0.8406, Log Rank; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.538 to 2.140]
Statistical Analysis 2: Comparison: Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 vs Randomization Phase: Pemetrexed 500 mg/m2; Test type: Superiority or Other; p = 0.3960, Log Rank; Hazard Ratio (HR) = 1.081, 95% CI 2-sided [0.599 to 1.949]

4. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response was measured from the time measurement criteria were met for CR or PR (whichever was first recorded) until the first date that recurrent or progressive disease (PD) was objectively documented (taking as reference for PD the smallest measurements recorded since treatment began). The duration of overall CR was measured from the time measurement criteria were first met for CR until the first date that recurrent disease was objectively documented. Duration of disease control is presented here.
Time Frame: From the time measurement criteria were met for CR or PR (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented
Population: Randomized phase II set
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Number analyzed (Participants) | 10 | 31 | 32
weeks | 23.0 [12.7 to 47.1] | 19.6 [7.1 to 39.1] | 23.4 [10.5 to 45.9]

5. Secondary Outcome: Occurrence and Intensity of AEs Graded According to CTCAE.
Description: All patients were carefully monitored during and after each treatment cycle. Adverse events (AEs) were recorded and were graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: From first drug infusion until 21 days after last drug infusion, up to 1100 days
Population: Treated set, which included all patients who were dispensed and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Number analyzed (Participants) | 6 | 6 | 36 | 46 | 46
participants
  CTCAE Grade 1 | 0 | 0 | 6 | 2 | 6
  CTCAE Grade 2 | 0 | 2 | 12 | 18 | 18
  CTCAE Grade 3 | 3 | 3 | 8 | 19 | 15
  CTCAE Grade 4 | 3 | 1 | 6 | 5 | 5
  CTCAE Grade 5 | 0 | 0 | 3 | 2 | 0

6. Secondary Outcome: Occurence of DLT
Description: Occurence of Dose-limiting toxicity (DLT). A DLT was defined as one or more of the following:
  * treatment-related CTCAE Grade 3 or 4 nonhematological toxicity (except emesis or diarrhea responding to supportive treatment).
  * treatment-related CTCAE Grade 4 neutropenia for ≥7 days and/or complicated by infection.
  * CTCAE Grade 4 thrombocytopenia.
Time Frame: Patients were treated for repeated 21-day treatment cycles until disease progression or intolerability of the trial drug, whichever occurred first.
Population: Treated set, run-in phase, first course only
Measure: Number; unit: participants
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2
Number analyzed (Participants) | 6 | 6
participants | 1 | 1

7. Secondary Outcome: Frequency of Patients With Possible Clinically Significant Abnormalities
Description: Frequency of patients with possible clinically significant abnormalities
Time Frame: From first drug infusion until 21 days after last drug infusion, up to 1100 days
Population: On-treatment for lab
Measure: Number; unit: participants
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Number analyzed (Participants) | 6 | 6 | 36 | 46 | 46
participants
  Haemoglobin - Low | 1 | 2 | 16 | 21 | 14
  White blood cell ct. - Low | 4 | 2 | 15 | 25 | 12
  White blood cell ct. - High | 0 | 0 | 1 | 0 | 1
  Platelets - Low | 0 | 1 | 8 | 3 | 2
  Platelets - High | 0 | 1 | 3 | 0 | 3
  Neutrophils - Low | 4 | 2 | 13 | 23 | 12
  Lymphocytes - Low | 4 | 4 | 16 | 22 | 22
  AST/GOT, SGOT - High | 0 | 1 | 0 | 6 | 3
  ALT/GPT, SGPT - High | 0 | 1 | 0 | 10 | 6
  Alkaline phosphatase - High | 0 | 0 | 0 | 0 | 5
  Creatinine - High | 0 | 0 | 0 | 3 | 0
  Bilirubin, total - High | 1 | 0 | 1 | 1 | 1

8. Secondary Outcome: Cmax of Volasertib
Description: Cmax - maximum measured concentration of volasertib in plasma.
Time Frame: 5 minutes (min) before the start of Volasertib infusion and 1 hour (h), 2h, 4h, 24h, 168h and 336h after the start of Volasertib infusion
Population: Pharmacokinetic (PK) set, which included all patients in the treated set with volasertib monotherapy or combined with pemetrexed and provided at least 1 blood sample for measurement of volasertib (BI 6727) or pemetrexed. Including patients with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Volasertib 250 mg + Pemetrexed 500 mg/m2: Patients received Volasertib 250 mg and pemetrexed 500 mg/m2 administered intravenously (i.v.) on day 1 of each 21 day cycle.
- Volasertib 300 mg + Pemetrexed 500 mg/m2: Patients received Volasertib 300 mg and pemetrexed 500 mg/m2 administered intravenously (i.v.) on day 1 of each 21 day cycle
- Volasertib 300 mg: Patient received Volasertib 300 mg administered intravenously on day 1 of each 21 day cycle.
Arm/Group | Volasertib 250 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg
Number analyzed (Participants) | 4 | 39 | 30
ng/mL | 554 (35.9) | 635 (51.8) | 565 (39.0)

9. Secondary Outcome: Total Clearance (CL) of Volasertib
Description: CL - total clearance of volasertib in plasma after IV administration
Time Frame: as for outcome 8
Population: PK set including patients with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Volasertib 250 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg
Number analyzed (Participants) | 6 | 46 | 30
mL/min | 782 (24.8) | 882 (30.4) | 867 (31.6)

10. Secondary Outcome: Vss of Volasertib
Description: Vss - apparent volume of distribution at steady state following IV administration of volasertib
Time Frame: as for outcome 8
Population: PK set including patients with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | Volasertib 250 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg
Number analyzed (Participants) | 6 | 46 | 30
Litres | 6730 (42.1) | 6750 (39.7) | 6230 (34.5)

11. Secondary Outcome: Cmax of Pemetrexed
Description: Cmax - maximum measured concentration of pemetrexed in plasma
Time Frame: 5 minutes before pemetrexed infusion, at the end of the infusion and 1.5 hours (h), 2.5h, 4.5h and 25.5h after the end of pemetrexed infusion
Population: PK set including patients with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Volasertib 250 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg + Pemetrexed 500 mg/m2
Number analyzed (Participants) | 6 | 38
ng/mL | 131000 (24.7) | 115000 (32.1)

12. Secondary Outcome: CL of Pemetrexed
Description: CL - total clearance of pemetrexed in plasma after IV administration
Time Frame: as for outcome 11
Population: PK set including patients with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Volasertib 250 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg + Pemetrexed 500 mg/m2
Number analyzed (Participants) | 5 | 43
mL/min | 54.4 (17.4) | 69.1 (30.0)

13. Secondary Outcome: Vss of Pemetrexed
Description: Vss - apparent volume of distribution at steady state following IV administration of pemetrexed
Time Frame: as for outcome 11
Population: PK set including patients with evaluable data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | Volasertib 250 mg + Pemetrexed 500 mg/m2 | Volasertib 300 mg + Pemetrexed 500 mg/m2
Number analyzed (Participants) | 5 | 43
Litres | 9.40 (20.5) | 13.1 (45.8)

ADVERSE EVENTS:
Time Frame: From first drug infusion until 21 days after last drug infusion, up to 1100 days
Arm/Group | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Volasertib 300 mg | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 | Randomization Phase: Pemetrexed 500 mg/m2
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 8/36 | 10/46 | 12/46
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 35/36 | 46/46 | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 (N=6) | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 (N=6) | Randomization Phase: Volasertib 300 mg (N=36) | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 (N=46) | Randomization Phase: Pemetrexed 500 mg/m2 (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Phase: Volasertib 250 mg + Pemetrexed 500 mg/m2 (N=6) | Run-in Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 (N=6) | Randomization Phase: Volasertib 300 mg (N=36) | Randomization Phase: Volasertib 300 mg + Pemetrexed 500 mg/m2 (N=46) | Randomization Phase: Pemetrexed 500 mg/m2 (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 12 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 9 | 9 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 4 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 2 | 3 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 3 | 0 | 0 | 2
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 2
Eye oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 1 | 7 | 7
Vision blurred (Eye disorders) | 1 | 1 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 6 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 6 | 17 | 10
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 4 | 14 | 12
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3 | 5 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 5 | 22 | 25
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 7 | 15 | 11
Asthenia (General disorders) | 0 | 2 | 4 | 2 | 1
Catheter site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 3 | 4 | 7 | 5
Chills (General disorders) | 0 | 0 | 3 | 4 | 2
Fatigue (General disorders) | 5 | 6 | 20 | 33 | 32
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 8 | 4
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 4 | 13 | 5
Pain (General disorders) | 0 | 0 | 3 | 4 | 3
Puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 3 | 7 | 9
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 4 | 3 | 8
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 3 | 5
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 3
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 2 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 9 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Carbohydrate antigen 125 increased (Investigations) | 1 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0 | 3 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 1 | 1 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 3 | 1 | 0
Weight decreased (Investigations) | 2 | 1 | 1 | 5 | 4
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 2 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 3 | 20 | 19
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 2
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 12 | 13 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 5 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5 | 5 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2 | 4
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 7 | 9 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 8 | 1
Headache (Nervous system disorders) | 0 | 2 | 2 | 9 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 3 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 5 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 3 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 4 | 7
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 2 | 3
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 4 | 4
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 9 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6 | 12 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 4 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 3 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 14 | 12
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 3 | 3
Hypertension (Vascular disorders) | 2 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.